CLINICAL TRIAL: NCT05007912
Title: Prospective Observational Study Comparing the Use of Circular (Orvil) and Linear Stapler for Intracorporeal Esophagojejunostomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH_EJ
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orvil Group: Group that used the Orvil (circular stapler) for esophagojejunostomy
  Interventions: Procedure: Esophagojejunostomy type
- Linear Group: Group that used the linear stapler for esophagojejunostomy
  Interventions: Procedure: Esophagojejunostomy type

INTERVENTIONS:
Procedure: Esophagojejunostomy type — Use of either circular or linear stapler

SUMMARY:
Prospective observational study comparing the use of circular (Orvil) and linear stapler for intracorporeal esophagojejunostomy.

Patients with adenocaricinoma involving the esophagogastric junction or the gastric cardia are observed. The two methods of esophagojejunostomy are compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as gastric adenocarcinoma
* Involving the esophagogastric junction or gastric cardia
* Age 18 - 80 years
* Anticipated to undergo laparoscopic total or proximal gastrectomy
* cT1-T4a

Exclusion Criteria:

* Previous history of gastrectomy
* Neoadjuvant chemotherapy or radiotherapy for gastric cancer
* Invasion to other organs
* Open conversion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients involving the upper stomach
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Anastomosis complication | within 1 year
  including anastomosis leakage, stenosis, bleeding of the esophagojejunostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No